CLINICAL TRIAL: NCT02751528
Title: Phase I Study of Ad5 [E1-, E2b-]-HER2/Neu Vaccine (ETBX-021) in Subjects With Unresectable Locally Advanced or Metastatic HER2-Low-Expressing (IHC 1+/2+) Breast Cancer
Brief Title: QUILT-3.013: Study of Ad5 [E1-, E2b-]-HER2/Neu Vaccine (ETBX-021) in Subjects With Unresectable Locally Advanced or Metastatic HER2-Expressing Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to low enrollment
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.013
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Breast Cancer; Breast Cancer male; Breast Neoplasms; Breast Neoplasms male; Vaccine; HER2; Metastatic; Locally Advanced; Unresectable; Solid Tumor; Phase 1; Cancer Vaccine
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Breast Neoplasms, Male; Neoplasm Metastasis | interventions — Presenilin-1; methyl N-acetylsibirosaminide; Suspensions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ETBX-021 (Experimental): Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection
  Interventions: Biological: ETBX-021

INTERVENTIONS:
Biological: ETBX-021 — ETBX-021 is a HER2-targeting vaccine comprising an Ad5 vector and a modified HER2 gene insert.
  Other Names: Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection

SUMMARY:
The purpose of this study is to determine whether ETBX-021 is safe and effective in the treatment of unresectable locally advanced or metastatic HER2-low-expressing breast cancer.

DETAILED DESCRIPTION:
This is a Phase I trial in subjects with unresectable locally advanced or metastatic HER2-low expressing (IHC 1+ or 2+) breast cancer. The study will be conducted in two parts: the first part will involve dose escalation using a 3 + 3 design, and the second part will involve the expansion of the MTD or HTD to further evaluate safety, preliminary efficacy, and immunogenicity. In the first part, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1. Subjects will be assessed for dose-limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Male or female.
3. Ability to understand and provide signed informed consent that fulfills Institutional Review Board (IRB)'s guidelines.
4. Histologically confirmed unresectable locally advanced or metastatic breast cancer that expresses HER2 (IHC 1+ or 2+), derived from the most recent metastatic biopsy sample available.
5. Tumor tissue (block or slides) and whole blood sample available for analysis. Archival tissue is permitted.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Concurrent hormone therapy is permitted.
8. Subjects who have received prior HER2-targeted immunotherapy (vaccine) are eligible for this trial if this treatment was discontinued at least 3 months prior to enrollment.
9. Resolution of all toxic side effects of prior chemotherapy, radiotherapy, or surgical procedures to NCI CTCAE Grade ≤ 1.
10. Subjects who are taking medications that do not have a known history of immunosuppression are eligible for this trial.
11. Adequate hematologic function at screening, as follows:

    * White blood count ≥ 3000/microliter.
    * Hemoglobin ≥ 9 g/dL (may not transfuse or use erythropoietin to achieve this level).
    * Platelets ≥ 75,000/microliter.
    * Prothrombin (PT)-international normalized ratio (INR) < 1.5.
    * Partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN).
12. Adequate renal and hepatic function at screening, as follows:

    * Serum creatinine < 2.0 mg/dL.
    * Bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL).
    * Alanine aminotransferase (ALT) ≤ 2.5 x ULN.
    * Aspartate aminotransferase (AST) ≤ 2.5 x ULN.
13. Multigated acquisition (MUGA) scan or echocardiogram with LVEF ≥ institutional LLN. Same imaging modality is to be used throughout the study.
14. Female subjects of childbearing potential and women < 12 months since the onset of menopause must agree to use acceptable contraceptive methods for the duration of the study and for 7 months following the last injection of study medication. If employing contraception, two of the following precautions must be used: vasectomy of partner, tubal ligation, vaginal diaphragm, intrauterine device, condom and spermicidal (gel/foam/cream/vaginal suppository), or total abstinence. Male subjects must be surgically sterile or must agree to use a condom and acceptable contraceptive method with their partner. Female subjects who are post-menopausal are defined as those with an absence of menses for > 12 consecutive months.
15. Ability to attend required study visits and return for adequate follow up, as required by this protocol.

Exclusion Criteria:

1. Subjects with HER2 IHC 3+ tumors, or IHC 2+ with an in situ hybridization (ISH) test result considered positive of HER2 amplification by ASCO-CAP HER2 test guidelines.
2. Subjects with ongoing HER2-directed therapy, including trastuzumab, pertuzumab, T-DM1, and lapatinib.
3. Participation in an investigational drug or device study within 30 days of screening for this study.
4. Pregnant and nursing women.
5. Subjects with ongoing palbociclib, everolimus, or other breast cancer therapy that interferes with the induction of immune responses.
6. Subjects with concurrent cytotoxic chemotherapy or radiation therapy. There must be at least 1 month between any other prior chemotherapy (or radiotherapy) and study treatment. Any prior HER2-targeted immunotherapy (vaccine) must have been discontinued at least 3 months before initiation of study treatment. Subjects must have recovered from all acute toxicities from prior treatment prior to screening for this study.
7. Active brain or central nervous system metastasis, seizures requiring anticonvulsant treatment, cerebrovascular accident (< 6 months), or transient ischemic attack.
8. Subjects with a history of autoimmune disease (active or past), such as but not restricted to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune-related thyroid disease and vitiligo are permitted.
9. Subjects with serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, or other illness considered by the Investigator as high risk for investigational drug treatment.
10. Subjects with a history of heart disease, such as congestive heart failure (class II, III, or IV defined by the New York Heart Association functional classification), history of unstable or poorly controlled angina, or history (< 1 year) of ventricular arrhythmia.
11. Subjects with a medical or psychological impediment that would impair the ability of the subject to receive therapy per protocol or impact ability to comply with the protocol or protocol-required visits and procedures.
12. History of malignancy except for the following: adequately treated non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other carcinoma that has been in complete remission without treatment for more than 5 years.
13. Presence of a known active acute or chronic infection, including human immunodeficiency virus (HIV, as determined by enzyme-linked immunosorbent assay [ELISA] and confirmed by western blot) and hepatitis B and hepatitis C virus (HBV/HCV, as determined by HBsAg and hepatitis C serology).
14. Subjects on systemic intravenous or oral steroid therapy (or other immunosuppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Subjects must have had at least 6 weeks of discontinuation of any steroid therapy (except that used as premedication for chemotherapy or contrast-enhanced studies) prior to enrollment.
15. Subjects with known allergy or hypersensitivity to any component of the investigational product will be excluded.
16. Subjects with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
17. Subjects vaccinated with a live (attenuated) vaccine (e.g., FluMist®) or a killed (inactivated)/subunit vaccine (e.g., PNEUMOVAX®, Fluzone®) within 28 days or 14 days, respectively, of the first planned dose of ETBX-021.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chan Soon-Shiong Institute for Medicine, El Segundo, California
  - Sanford Cancer Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 x 10^10 VP: Ad5 [E1-, E2b-]-HER2/neu Vaccine, Suspension for Injection
  ETBX-021: ETBX-021 is a HER2-targeting vaccine comprising an Ad5 vector and a modified HER2 gene insert.
Period: Overall Study
Arm/Group | 5 x 10^10 VP
Started | 3
Completed | 1
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (3.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Histologically confirmed unresectable locally advanced or metastatic breast cancer that expresses HE [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events, Number of Participants With Treatment Emergent Serious Adverse Events, and Number of Participants With Dose Limiting Toxicities (DLTs)
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Participants
  TEAE | 3
  TESAE | 1
  DLT | 0

2. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) or Highest Tested Dose (HTD)
Time Frame: Up to 11 months
Population: MTD / HTD not reached due to early termination of the study
Measure: Number; unit: virus particles
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
virus particles | NA — MTD / HTD not reached due to early termination of the study

3. Secondary Outcome: ORR (Confirmed Complete or Partial Response)
Description: ORR assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Time Frame: Up to 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | ETBX-021
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Confirmed response or stable disease lasting for at least 6 months according to RECIST V1.1
Time Frame: Up to 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Participants | 1

5. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrence or PD is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: Up to 11 months
Population: Best overall response was Stable Disease, which did not meet the criteria for duration of response.
Measure: Number; unit: Months
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Months | NA — Best overall response was Stable Disease, which did not meet the criteria for duration of response.

6. Secondary Outcome: Progression Disease Survival
Description: PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurred first.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Months | NA [1.7 to NA] — N/A - Median time and upper limit of 95% CI were not reached.

7. Secondary Outcome: Overall Survival
Description: OS will be defined as the time from the date of first treatment to the date of death (any cause).
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 5 x 10^10 VP
Number analyzed (Participants) | 3
Months | NA [1.7 to NA] — N/A - Median time and upper limit of 95% CI were not reached.

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of the study drug, up to 12 months. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 12 months. All SAEs that have not resolved upon discontinuation of the subject's participation in the study must be followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow up, or otherwise explained, up to 12 months.
Arm/Group | 5 x 10^10 VP
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 x 10^10 VP (N=3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 x 10^10 VP (N=3)
Injection site reaction (General disorders) | 2
Pyrexia (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral dysaesthesia (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT02751528/Prot_SAP_000.pdf